CLINICAL TRIAL: NCT01520493
Title: Peripheral Muscle Microcirculation and Exercise-induced Blood Flow Distribution in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Steeve Provencher, Professeur, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Microcirculation_Local funds
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; skeletal muscle microcirculation; exercise induced blood flow
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): All patients are subject to this Arm.
  Interventions: Other: Submaximal exercises

INTERVENTIONS:
Other: Submaximal exercises — Consists of a 3-min unloaded exercise, followed by a progressive RAMP protocol (10 watts/min) up to 70% of peak workload followed by 3 min. of cycling at constant workload (70% peak workload) (total exercise duration of 25 min.).

SUMMARY:
Pulmonary artery hypertension (PAH) is a rare, severe disease, characterized by a progressive increase in pulmonary vascular resistance ultimately leading to right ventricular (RV) failure and premature death. PAH may be idiopathic (IPAH) or may be also related to various conditions like portal hypertension, HIV infection, left to right shunt, connective tissue diseases such as scleroderma (PAHSSc). Symptoms include dyspnea and fatigue resulting in restricted exercise capacity and poor quality of life. The therapies currently approved have been shown to improve survival. Indeed, recent studies described a three year survival higher than 80%. This improved survival is associated with major challenges for clinicians as most patients remain with limited exercise capacity and poor quality of life. A clear understanding of exercise physiopathology is thus mandatory to specifically address mechanisms responsible for this exercise limitation and eventually improve patients' management. In order to better characterize the exercise physiopathology in PAH, the general objective of this research is to systematically examine blood flow distribution and limb muscles microcirculation at rest and during submaximal exercise in PAH.

DETAILED DESCRIPTION:
Pulmonary artery hypertension (PAH) is a rare, severe disease, characterized by a progressive increase in pulmonary vascular resistance ultimately leading to right ventricular (RV) failure and premature death. PAH may be idiopathic (IPAH) or may be also related to various conditions like portal hypertension, HIV infection, left to right shunt, connective tissue diseases such as scleroderma (PAHSSc). PAH is defined as a mean pulmonary artery pressure (mPAP) of > 25 mmHg at rest. Symptoms include dyspnea and fatigue resulting in restricted exercise capacity and poor quality of life. The agents currently approved for treatment of PAH are prostanoids (i.v. epoprostenol or s.c./i.v. treprostinil), endothelin-receptor antagonists (ambrisentan, bosentan and sitaxsentan), and phosphodiesterase type 5-inhibitors (sildenafil and tadalafil). These therapies have been shown to improve pulmonary hemodynamics, exercise capacity, quality of life and survival. Indeed, recent studies described a three year survival higher than 80%. This improved survival is associated with major challenges for clinicians as most patients remain with limited exercise capacity and poor quality of life. A clear understanding of exercise physiopathology is thus mandatory to specifically address mechanisms responsible for this exercise limitation and eventually improve patients' management.

In order to better characterize the exercise physiopathology in PAH, the general objective of this research is to systematically examine blood flow distribution and limb muscles microcirculation at rest and during submaximal exercise in PAH. The limited link between traditional measures of pulmonary hemodynamic impairment and functional capacity confirms that exercise physiopathology in PAH is not well understood. Although peripheral muscle dysfunction and exercise intolerance are certainly multifactorial in origin and are unlikely to be explained by a single mechanism, an altered skeletal muscle microcirculation could represent a unifying mechanism to explain similarities in skeletal muscle dysfunction and exercise intolerance in PAH. The investigators plan to use a multimodality approach to provide comprehensive information regarding skeletal muscle perfusion in PAH. For example, the investigators will be able to know if there is some relationship between muscle perfusion heterogeneity (arterial spin labeling MRI) and microvascular oxygenation or muscle oxygen consumption (NIRS). Muscle oxygen delivery could also be influenced by cardiac function or hypoxemia. These methods should thus be viewed as complimentary and will help to separate differences in cardiac function, quadriceps global perfusion, perfusion heterogeneity and oxygenation and their consequences on skeletal muscle function and exercise tolerance in PAH versus controls.

ELIGIBILITY:
Inclusion Criteria:

* WHO functional class II-III idiopathic PAH patients;
* WHO functional class II-III PAH-SSc patients with hemodynamic assessment <6 months;
* sedentary healthy subjects;
* subjects with limited SSc (without PAH) individually matched for age, gender, height and weight.

Exclusion Criteria:

1. unstable clinical condition (e.g. recent syncope, WHO functional class IV);
2. a six-minute walked distance < 300 meters during routine follow-up at the pulmonary hypertension clinic;
3. left ventricular ejection fraction < 40%;
4. restrictive (lung fibrosis on CT scan or total lung capacity < 80% of predicted) or obstructive lung disease (FEV1/FVC < 70%);
5. contraindication for MRI;
6. body mass index > 30 kg/m2;
7. known locomotor abnormality.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Muscle microcirculation during submaximal exercise | day 3
  Thigh muscles overall perfusion and perfusion heterogeneity will be assessed by pulsed arterial spin labeling magnetic resonance imaging (ASL MRI). MRI allows the acquisition of both spatially and temporally localized perfusion measurements within working muscle.
Cardiac output during submaximal exercise | day 3
  Cardiac MRI. Right after muscles perfusion heterogeneity assessment by MRI (both at rest and following the same exercise protocol), cardiac MRI will be performed with the same 1.5 Tesla MRI.
Muscle sympathetic nerve activity (MSNA) | day 2
  MSNA will be assessed by microneurography and measures sympathetic nerve traffic directed to muscle circulation. All measurements will be performed under quiet resting supine conditions before non-MRI exercise.
Quadriceps muscle function | day 2
  Quadriceps muscle function will be assessed using voluntary and non-volitional measurements:
  Strength of the dominant quadriceps will be evaluated using the Biodex System 4 Pro (Biodex Medical Systems, 20 Ramsay Road, Shirley, New York).
  Non-volitional dominant quadriceps endurance will be evaluated by magnetic stimulation of the femoral nerve using the Magstim Rapid 2 system (Magstim Co. Ltd., Whitland, Dyfed, Wales, UK) coupled with the Biodex System 4 Pro, allowing measurements of intrinsic muscle endurance properties independent of central drive.
Relationship between in vivo muscle microcirculation and capillarity | day 1
  Capillarity and angiogenesis-related gene expression in muscle biopsy. In order to explore the relationship between in vivo muscle microcirculation and capillarity, percutaneous biopsy specimens of the vastus lateralis muscle of the nondominant leg will be taken at midthigh as described by Bergström.

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, MSc, Principal Investigator — Fondation IUCPQ
Locations (2):
- Canada (2):
  - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec